CLINICAL TRIAL: NCT06272604
Title: Personalized Exercise Rehabilitation for Pediatric and Adolescent Asthma: A Comprehensive Intervention Study
Brief Title: Exercise Rehabilitation for Children With Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Nan Lin, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-IRB-0015-P-01
Record Dates: First submitted 2024-01-31; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Asthma in Children; Rehabilitation; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention Control Group (No Intervention): The control group will not receive any specific intervention, continuing with their usual asthma management routine.
- Exercise Rehabilitation Group (Experimental): The experimental group will participate in a 12-week exercise intervention program.
  Interventions: Behavioral: Personalized Exercise Rehabilitation

INTERVENTIONS:
Behavioral: Personalized Exercise Rehabilitation — The experimental group will participate in a 12-week exercise intervention program, carefully transitioning from moderate-intensity interval training to high-intensity interval training. The progression of exercise intensity will be regularly adjusted based on each child's tolerance, ensuring a personalized approach to the regimen. The exercise program is structured into three phases: an adaptation phase, an intensification phase, and a consolidation phase. For each participant, the intensity of the exercises is calculated based on their reserve heart rate, allowing for a tailored and scientifically-grounded progression. This approach aims to optimize the exercise program's effectiveness while maintaining safety and adaptability to individual fitness levels and asthma conditions.
  Arms: Exercise Rehabilitation Group

SUMMARY:
Asthma, a prevalent chronic condition among children and adolescents, substantially impairs their quality of life. In addressing this significant health concern, this study focuses on the potential of a customized exercise rehabilitation program tailored for this young demographic. By employing a randomized controlled trial design, the research aims to divide participants into two distinct groups: one undergoing a personalized exercise regimen and the other receiving standard medical care. The 12-week intervention for the exercise group includes a combination of aerobic activities, strength training, and targeted breathing exercises. The study's primary aim is to rigorously evaluate the impact of this specialized exercise protocol on critical health aspects such as lung function, physical endurance, frequency of asthma attacks, and overall quality of life. The anticipated findings from this research are expected to shed new light on effective asthma management strategies and offer invaluable guidance for clinical practices dedicated to improving health outcomes in young asthma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with bronchial asthma;
2. No acute asthma attacks in the past three months;
3. Currently undergoing stable prophylactic treatment for asthma, with no changes in the treatment plan in the past three months.

Exclusion Criteria:

1. Suffering from other severe heart, lung, or musculoskeletal diseases;
2. Frequent acute asthma attacks or recent hospitalization records;
3. Changes in asthma medication treatment plan in the last three months;
4. Currently participating in other clinical trials that could affect the results of this study;
5. Any medical contraindications, such as severe exercise-induced asthma or other health issues affecting the ability to exercise;
6. Severe psychological or behavioral issues that may affect participation in training or adherence to the research protocol.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Lung Function | up to 24 weeks
  Forced Vital Capacity (FVC), Forced Expiratory Volume in One Second (FEV1), Forced Expiratory Flow 25% to 75% (FEF25-75), Peak Expiratory Flow (PEF)
Daily Physical Activity Level | up to 24 weeks
  Daily Step Count (as measured by a pedometer), Energy Expenditure,Time Spent in Moderate-to-Vigorous Intensity Activity

SECONDARY OUTCOMES:
Asthma Control Status | up to 24 weeks
  asthma control test(ACT)
Fractional Exhaled Nitric Oxide (FeNO) | up to 12 weeks
  FeNO was determined by NIOX VERO
Body Composition | up to 24 weeks
  Height, Weight, Body Fat, Skeletal Muscle Content
Sleep | up to 24 weeks
  Number of Nighttime Awakenings, Sleep Duration
Health Related Quality of Life | up to 24 weeks
  Asthma Quality of Life Questionnaire
Anxiety and Depression | up to 24 weeks
  C-C-Ped-PROMIS
Inflammatory Mediators | up to 12 weeks
  IL-4, IL-5, IL-13